CLINICAL TRIAL: NCT00983970
Title: Effects of Interactive Video Game Cycling on Obese Adolescent Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Dr. Gary Goldfield, Senior Scientist, Children's Hospital of Eastern Ontario Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-2-06-2106-GG; CDA-GG-2-06-2106-GG
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Overweight With Comorbidity; Obesity
Keywords: Adolescents; Obesity; Exercise; Music; Virtual Reality
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive video cycling (Experimental): Interactive video cycling arm utilized the Gamebike that interfaced a Sony Play Station 2 with a stationary bicycle and a 42 inch flat screen TV. The Gamebike has a handle bar mounted game controller allowing the participant to play most Sony Play Station 2 raced-based video games. The Gamebike reads the participants' speed by cycling cadence and the faster the individual pedalled, the faster they moved in the virtual world on screen. Participants were asked to come to the lab for two sessions per week for 60 minutes for 10 weeks.Participants were told that they could exercise at any intensity or duration that they desired, and reading materials were provided for those who did not chose to exercise for the full 60 minute session.
  Interventions: Behavioral: Interactive video game cycling
- Cycling to Music (Active Comparator): Each participant exercised twice weekly for 10 weeks on the Gamebike® but the games and controls were turned off. The Gamebike® was used by both groups to control for any differences between two cycle ergometers such as comfort or usability. However, participants were allowed to listen to music of their choice via radio, CD or personal music device.
  Interventions: Behavioral: Cycling to Music

INTERVENTIONS:
Behavioral: Interactive video game cycling — Participants were required to exercise on a Gamebike® (Cat Eye Electronics Ltd, Boulder Col.) interactive video gaming system that was interfaced with a Sony Play Station 2® (Sony computer Entertainment America Inc. Foster, City, CA) and a 42" flat screen television monitor. The Gamebike® has a handlebar mounted game controller allowing the participant to play most Sony Playstation 2- race-based video games. The Gamebike® reads the participant's speed by cycling cadence and the faster the individual pedalled, the faster they moved in the virtual world on screen. Participants were told that they could exercise at any intensity and duration they desired. Participants were asked to come to the lab for two sessions per week for 60 minutes for 10 weeks. Although participants were required to stay in the lab for 60 minutes, they could take breaks or stop when they wanted, and reading materials were available for those who did not or could not cycle for the full 60 minute session.
  Arms: Interactive video cycling
Behavioral: Cycling to Music — Each participant exercised twice weekly for 10 weeks on the Gamebike® but the games and controls were turned off. The Gamebike® was used by both groups to control for any differences between two cycle ergometers such as comfort or usability. However, participants were allowed to listen to music of their choice via radio, CD or personal music device. We incorporated music into the control condition because most youth and young adults exercise to music and this provides a more stringent test of the Gamebike® while improving the ecological validity of the research design. We also wanted to minimize drop-out and felt that expecting overweight/obese adolescents, who often report disliking aerobic exercise, to bike in a lab with no form of distraction would create a less than desirable exercise environment and result in high drop-out rates.
  Arms: Cycling to Music

SUMMARY:
Exercise is an important component in the treatment of of child obesity and associated medical conditions. However, one of the strongest predictors of non-compliance from exercise programs in obese youth is lack of enjoyment, thus creating a more pleasurable environment, by using TV or video games as incentives, may be an effective way of increasing exercise in obese youth. The purpose of this study was to compare interactive video game stationary cycling (GameBike ®) with cycling to music on aerobic fitness, body composition, cardiovascular disease risk markers, and exercise behaviour as measured by attendance, energy expenditure, duration, intensity and distance pedaled in obese adolescents. Twenty six obese adolescents had an equal chance of being assigned to either interactive video game cycling (n=13) or cycling to music serving as controls (n=13). The 10-week program consisted of twice weekly sessions lasting a maximum of 60 minutes per session.

DETAILED DESCRIPTION:
Background: Energy expenditure through exercise is important for weight loss and reduction of medical morbidity associated with adolescent obesity. However, attrition from aerobic exercise programs is high in obese children as they do not tolerate it or enjoy it. Capitalizing on technology to use TV or video games as incentives to exercise may improve adherence to exercise and associated health benefits in obese adolescents.

Objective: The purpose of this study was to compare the efficacy of interactive video game stationary cycling (GameBike ®) with cycling to music on aerobic fitness, body composition, cardiovascular disease risk markers, and exercise behaviour as measured by attendance, energy expenditure, duration, intensity and distance pedaled in obese adolescents.

Method: Twenty six obese adolescents were stratified by gender and randomized to a either interactive video game cycling (n=13) or cycling to music serving as controls (n=13). The 10-week program consisted of twice weekly sessions lasting a maximum of 60 minutes per session.

ELIGIBILITY:
Inclusion Criteria:

* youth aged 12-17 years with BMI above 95th percentile for age and gender based on CDC growth chart data, OR
* BMI > 85th percentile for age and gender with one of the following:
* elevated fasting glucose or 2 hour OGTT (indicative of impaired glucose tolerance)
* elevated fasting triglycerides, LDL-C, reduced HDL-C
* total cholesterol/HDL-C ratio > 90th percentile
* elevated fasting insulin
* Blood pressure > 90th percentile
* 1st degree relative with Type II diabetes or cardiovascular disease
* Willingness to follow protocol and sign informed assent and consent

Exclusion Criteria:

* Did not have a medical condition that altered intestinal absorption
* Did not influence response to activity intervention or make vigorous exercise dangerous - such as
* type 1 diabetes mellitus
* inflammatory bowel disease,
* severe arthritis/asthma,
* congestive heart failure,
* pulmonary disease,
* systemic hypertension,
* acute renal disease
* other illness assessed by the study physician making participation inadvisable

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure (kilocalories) | baseline and 10-weeks

SECONDARY OUTCOMES:
Aerobic fitness | baseline and 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Goldfield, Ph.D., Principal Investigator — Children's Hospital of Eastern Ontario Research Institute; Kristi B Adamo, PhD., Principal Investigator — Children's Hospital of Eastern Ontario Research Institute; Jane A Rutherford, MSc, Study Director — Children's Hospital of Eastern Ontario Research Institute
Locations (1):
- Children's Hospital Of Eastern Ontario Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Thivel D, Chaput JP, Adamo KB, Goldfield GS. Is energy intake altered by a 10-week aerobic exercise intervention in obese adolescents? Physiol Behav. 2014 Aug;135:130-4. doi: 10.1016/j.physbeh.2014.06.013. Epub 2014 Jun 19. PMID 24952265